CLINICAL TRIAL: NCT00543010
Title: MK0767 Glipizide Comparator Cardiac Safety Study (0767-018)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-018; 2007_644
Record Dates: First submitted 2007-10-05; First posted 2007-10-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
A study to evaluate the cardiac and metabolic effects of MK0767 in patients with Type 2 Diabetes.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* You are taking at least one medication for high blood sugar
* Age 21 to 80

Exclusion Criteria:

* History of Type 1 Diabetes Mellitus
* Currently on estrogen replacement therapy regimen
* Currently on a weight loss program with ongoing weight loss or taking medications for weight loss
* Having surgery 30 days before starting the study
* Have taken any other investigational drug in the past 90 days
* Have Hepatitis B or C
* Active liver or gallbladder disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2002-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC